CLINICAL TRIAL: NCT01800942
Title: Prevention of Bacterial Infections in the Newborn by Pre-delivery Administration of Azithromycin (AZI): a Placebo-controlled Randomized Trial
Brief Title: Prevention of Bacterial Infections in Newborn
Acronym: PregnAnZI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCC1282
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Neonatal Infection
Keywords: prevention; bacterial infection; neonates; women in labour; Azithromycin
MeSH Terms: conditions — Bacterial Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 830 women will be recruited into the study and randomised in a ratio of 1:1 per study arm to receive either Azithromycin or placebo.
  A single dose of Azithromycin 2g or Placebo will be given orally to pregnant women in labour.
  Interventions: Drug: Azithromycin and Placebo
- Azithromycin (Experimental): 830 women will be recruited into the study and randomised in a ratio of 1:1 per study arm to receive either Azithromycin or placebo.
  A single dose of Azithromycin 2g or Placebo will be given orally to pregnant women in labour.
  Interventions: Drug: Azithromycin and Placebo

INTERVENTIONS:
Drug: Azithromycin and Placebo — A single oral dose of 2g of Azithromycin will be given to the women in labour

SUMMARY:
The last decade has witnessed an important reduction of the mortality in children under 5 years but such reduction has not impacted in neonates. Mortality in neonates contributes 40% of all deaths occurring in children below 5 years of age.

Severe bacterial disease is among the leading causes of neonatal deaths. Bacterial disease follows bacterial infection. Individuals can be infected without developing disease (carriage stage) but infection is needed to subsequently develop disease. In sub-Saharan Africa, bacterial carriage (i.e. in the birth canal and/or nasopharyngeal tract) is very common in all age groups, with the consequence that occurrence of bacterial disease is one of the highest in the world.

Newborns can be infected during labour - when passing through the birth canal - and during the first days/weeks of life, as a consequence of the close physical contact with the mother, if the latter carries bacteria in the nasopharyngeal tract.

If the mother is an important source of bacterial infection to the newborn, treating mothers with a powerful antibiotic during labour should decrease bacterial carriage and therefore diminish the risk of bacterial transmission to the newborn during the first days/weeks of life, which should in turn result in the lower occurrence of severe bacterial disease and hence lower mortality.

The purpose of this trial is to evaluate the impact of a single oral dose of azithromycin given to women in labour on bacterial carriage of the newborn as well as the women during the first month after delivery.

The investigators have selected an antibiotic (azithromycin) that in sub-Saharan Africa has already shown both a strong impact on bacterial nasopharyngeal carriage and on all-cause mortality when administered to everybody in a community (mass drug administration). This specific antibiotic has several advantages for being deployable as a simple intervention in rural Africa, i.e. it requires a single oral administration, it has no special storage requirements and it has the potential to eliminate many of the bacteria commonly causing severe disease in newborn.

This clinical trial will be conducted in a peri-urban health facility in Western Gambia. If an impact is shown, the next step would be to conduct a larger study aiming at establishing if the intervention, implemented at a lower level of care (most African women deliver at home assisted by traditional birth assistants), decreases the occurrence of neonatal bacterial disease

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (aged 18 to 45 years)
* in labour
* attending a health centre in western Gambia for delivery

Exclusion Criteria:

* Known HIV infection.
* Any chronic or acute conditions of the women that might interfere with the study as judged by the research clinician.
* Planned travelling out of the catchment area during the following 2 months (follow-up period)
* Planned caesarean section
* Known required referral
* Known multiple pregnancy
* Known severe congenital malformation
* Intrauterine death confirmed before randomization
* Known allergy to macrolides
* Consumption of antibiotic within the week before randomisation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 829 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
the prevalence of nasopharyngeal carriage of the newborn of any of the following bacteria: 1) Group B Streptococci (GBS) , 2) S.pneumoniae and 3) S.aureus | 6 days
  The primary outcome is the prevalence of nasopharyngeal carriage of the newborn at the age of six days for any of the following bacteria: 1) Group B Streptococci, 2) S.pneumoniae and 3) S.aureus.

SECONDARY OUTCOMES:
Vaginal bacterial Group B Streptococci(GBS), S.pneumoniae and S.aureus) carriage at day six post-delivery. Vaginal bacterial (GBS, S.pneumoniae and S.aureus) carriage at day 8-10 post-delivery | 6-13 days
  The secondary outcomes are the prevalence of:
  - Newborn's nasopharyngeal bacterial Group B Streptococci (GBS), S.pneumoniae and S.aureus) carriage at any other scheduled visit.
  Bacterial isolates Group B Streptococci (GBS), S.pneumoniae and S.aureus), both from the newborn and the mother, non-susceptible to macrolides, from different study samples and time-points.
  Bacterial Group B Streptococci (GBS), S.pneumoniae and S.aureus) carriage in the breast milk at any scheduled visit.
  Purulent conjunctivitis within the first 4 weeks of life. Purulent Chlamydial conjunctivitis. AZI levels in breast milk on day 3 and 6 post-delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Roca, PhD, Principal Investigator — Medical Research Council Unit, The Gambia
Locations (1):
- Medical Research Council Unit, Fajara, The Gambia

REFERENCES:
- [Derived] Jagne I, Keeley AJ, Bojang A, Camara B, Jallow E, Senghore E, Oluwalana C, Bah SY, Turner CE, Sesay AK, D'Alessandro U, Bottomley C, de Silva TI, Roca A. Impact of intra-partum azithromycin on carriage of group A streptococcus in the Gambia: a posthoc analysis of a double-blind randomized placebo-controlled trial. BMC Infect Dis. 2022 Jan 29;22(1):103. doi: 10.1186/s12879-022-07080-4. PMID 35093029
- [Derived] Camara B, Oluwalana C, Miyahara R, Lush A, Kampmann B, Manneh K, Okomo U, D'Alessandro U, Roca A. Stillbirths, Neonatal Morbidity, and Mortality in Health-Facility Deliveries in Urban Gambia. Front Pediatr. 2021 Feb 15;9:579922. doi: 10.3389/fped.2021.579922. eCollection 2021. PMID 33659227
- [Derived] Bojang A, Baines SL, Camara B, Guerillot R, Donovan L, Marques RS, Secka O, D'Alessandro U, Bottomley C, Howden BP, Roca A. Impact of Intrapartum Oral Azithromycin on the Acquired Macrolide Resistome of Infants' Nasopharynx: A Randomized Controlled Trial. Clin Infect Dis. 2020 Dec 15;71(12):3222-3225. doi: 10.1093/cid/ciaa609. PMID 32445474
- [Derived] Bojang A, Baines SL, Donovan L, Guerillot R, Stevens K, Higgs C, Bottomley C, Secka O, Schultz MB, Goncalves da Silva A, Seemann T, Stinear TP, Roca A, Howden BP. Genomic investigation of Staphylococcus aureus recovered from Gambian women and newborns following an oral dose of intra-partum azithromycin. J Antimicrob Chemother. 2019 Nov 1;74(11):3170-3178. doi: 10.1093/jac/dkz341. PMID 31424550
- [Derived] Roca A, Camara B, Oluwalana C, Lette K, Bottomley C, D'Alessandro U. Long-lasting effect of oral azithromycin taken by women during labour on infant nutrition: Follow-up cohort of a randomized clinical trial in western Gambia. PLoS One. 2018 Oct 25;13(10):e0206348. doi: 10.1371/journal.pone.0206348. eCollection 2018. PMID 30359447
- [Derived] Bojang A, Camara B, Jagne Cox I, Oluwalana C, Lette K, Usuf E, Bottomley C, Howden BP, D'Alessandro U, Roca A. Long-term Impact of Oral Azithromycin Taken by Gambian Women During Labor on Prevalence and Antibiotic Susceptibility of Streptococcus pneumoniae and Staphylococcus aureus in Their Infants: Follow-up of a Randomized Clinical Trial. Clin Infect Dis. 2018 Sep 28;67(8):1191-1197. doi: 10.1093/cid/ciy254. PMID 29608659
- [Derived] Burr SE, Camara B, Oluwalana C, Bojang E, Bottomley C, Bojang A, Bailey RL, D'Alessandro U, Roca A. Does azithromycin given to women in labour decrease ocular bacterial infection in neonates? A double-blind, randomized trial. BMC Infect Dis. 2017 Dec 28;17(1):799. doi: 10.1186/s12879-017-2909-4. PMID 29282015
- [Derived] Roca A, Oluwalana C, Bojang A, Camara B, Kampmann B, Bailey R, Demba A, Bottomley C, D'Alessandro U. Oral azithromycin given during labour decreases bacterial carriage in the mothers and their offspring: a double-blind randomized trial. Clin Microbiol Infect. 2016 Jun;22(6):565.e1-9. doi: 10.1016/j.cmi.2016.03.005. Epub 2016 Mar 26. PMID 27026482
- [Derived] Salman S, Davis TM, Page-Sharp M, Camara B, Oluwalana C, Bojang A, D'Alessandro U, Roca A. Pharmacokinetics of Transfer of Azithromycin into the Breast Milk of African Mothers. Antimicrob Agents Chemother. 2015 Dec 28;60(3):1592-9. doi: 10.1128/AAC.02668-15. PMID 26711756
- [Derived] Roca A, Oluwalana C, Camara B, Bojang A, Burr S, Davis TM, Bailey R, Kampmann B, Mueller J, Bottomley C, D'Alessandro U. Prevention of bacterial infections in the newborn by pre-delivery administration of azithromycin: Study protocol of a randomized efficacy trial. BMC Pregnancy Childbirth. 2015 Nov 19;15:302. doi: 10.1186/s12884-015-0737-3. PMID 26585192